CLINICAL TRIAL: NCT07017296
Title: The In Vivo Anti-hypertensive Evaluation of Microencapsulated Pomegranate Juice Decreases the Diastolic Pressure in the Postprandial
Brief Title: Microencapsulated Pomegranate Juice as Anti-Hypertensive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma del Estado de Hidalgo (Other)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Gabriel Betanzos-Cabrera PhD, Researcher-Professor, Universidad Autónoma del Estado de Hidalgo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAEH-ICSA
Record Dates: First submitted 2025-05-20; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Clinical Trial
Keywords: hypertensive; microencapsulated pomegranate juice; fresh pomegranate juice
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: A group of twenty adult women from the "Ejido de Paraiso" health center, Sanitary Jurisdiction 2 Tulancingo de Bravo, Hidalgo Mexico,
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Water (Placebo Comparator): Water as placebo
  Interventions: Other: Placebo
- Positive control (Active Comparator): normal anti-hypertensive medication
  Interventions: Drug: Positive control
- Microencapsulated pomegranate juice (Experimental): treated with Microencapsulated pomegranate juice
  Interventions: Dietary Supplement: Active comparator
- Fresh pomegranate juice (Experimental): treated with fresh pomegranate juice
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Other: Placebo — 150 mL of water during the breakfast
  Arms: Water
Drug: Positive control — Normal antihypertensive in 150 ml of water during the breakfast
  Other Names: medication
  Arms: Positive control
Dietary Supplement: Active comparator — 20 g microencapsulated pomegranate juice in 150 mL water
  Arms: Microencapsulated pomegranate juice
Dietary Supplement: Control — 150 mL fresh pomegranate juice
  Arms: Fresh pomegranate juice

SUMMARY:
Introduction: Hypertension is a significant risk factor for cardiovascular disease (CVD). Pomegranate is a fruit rich in polyphenols that exerts an antihypertensive effect. Objective: The present work evaluated microencapsulated pomegranate juice (MPJ) as an anti-hypertensive in patients with mild hypertension. Materials and Methods: The content of phenols, flavonoids, anthocyanins, and antioxidant activity in fresh pomegranate juice (FPJ) and MPJ was determined. Subsequently, the postprandial anti-hypertensive effect was evaluated in recruited participants who consumed approximately 480 kcal breakfast. Four experimental groups with five participants each were evaluated: FPJ, 150 mL fresh juice; MPJ, 20 g microencapsulated pomegranate juice; the participant's usual drug (AH); and 150 mL water (W) with breakfast. Each participant's blood pressure (BP) was measured before and after breakfast at 30, 60, 90, and 120-min. Changes in BP values were evaluated as a function of time using generalized linear models.

DETAILED DESCRIPTION:
This study was conducted under the Law of General Health of Mexico, which was based on the 1964 Declaration of Helsinki. After a thorough review, the local Ethics Committee of Ministry of Health of Hidalgo approved the study (register number FSSA2021106). All participants signed a document indicating their informed consent. A group of twenty women from the "Ejido de Paraiso" Health Center, Sanitary Jurisdiction 2 Tulancingo de Bravo, Hidalgo México, were enrolled. Participation was based on the following inclusion criteria: patients fully diagnosed with mild hypertension values ranging from 140-159 mmHg/90-99 mmHg, and participants agreed to withhold anti-hypertensive medication for 48 h before the measurements. Participants' mean age was 56.31 ± 10.8 years. Women were selected for this study to avoid gender-bias which could result from a male and female cohort. In past decades, women have been under-represented in health care studies. Women allergic to the pomegranate fruit or diagnosed with COVID-19 were excluded.

The population was divided into four groups of 5 participants each as follows: 1) W, 150 mL of water; 2) AH, drug in 150 mL of water; 3) FPJ, 150 mL fresh pomegranate juice*; 4) MPJ, 20 g microencapsulated pomegranate juice in 150 mL water*. Asterisk (*) indicates an equivalent to 1.5 mmoles of total polyphenols. Breakfast consisted of two slices of whole wheat bread, two slices of turkey and pork ham, 30 g of panela cheese, one slice of tomato, one teaspoon of mayonnaise, two tablespoons of beans, and one cup of ultra-pasteurized whole milk.

Variables The dependent variable was arterial blood pressure (systolic or diastolic); measurements were taken in duplicate using a calibrated sphygmomanometer at pre-prandially (time 0) and post-prandially at 30, 60, 90, and 120 minutes after the meal. Time intervals were chosen to capture the immediate and short-term effects of the interventions on blood pressure.

The model was adjusted for two variables: Age in years, and Body Mass Index (BMI) in kg/m2. Estimation of BMI was based on Body weight in kilograms (kg) and height in meters (M). To estimate the changes in blood pressure in each period concerning time 0, 4 dummy variables with values of 0 or 1 were considered, for each postprandial period (at 30, 60, 90, and 120 minutes).

Participant data analysis Baseline measurements as mean ± standard deviation; an ANOVA test was used to assess differences between the study groups. Changes in blood pressure were evaluated using a generalized linear model (adjusted for BMI and age). The results of the model (coefficients) show the changes between each time point (30, 60, 90, and 120 minutes) relative to time 0 (baseline period) in mm/Hg. Statistical significance was defined as a p-value <0.05. All analyses were performed with the Statistical Program Package for the Social Sciences (SPSS) version 15 (SPSS, Inc., Chicago, Illinois USA).

ELIGIBILITY:
Inclusion Criteria:

* patients fully diagnosed with mild hypertension values ranging from 140-159 mmHg/90-99 mmHg
* participants agreed to withhold anti-hypertensive medication for 48 h before the measurements

Exclusion Criteria:

* Patients who were taking or were taking any product used as antihypertensive before 48h.
* Patients who were allergic to pomegranate fruit.
* Patients who did not attend a consultation at the health center.
* Patients diagnosed with Coronavirus disease 2019 (COVID-19).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics of the participants, overall and by study group | data collection at the beginning of the study, 10 days
  age in years
Baseline characteristics of the participants, overall and by study group | data collection at the beginning of the study, 10 days
  weight in kilograms
Baseline characteristics of the participants, overall and by study group | data collection at the beginning of the study, 10 days
  Height in meters
Baseline characteristics of the participants, overall and by study group | data collection at the beginning of the study, 10 days
  systolic and diastolic arterial pressure in mmHg

SECONDARY OUTCOMES:
Changes in systolic and diastolic blood pressure at different postprandial periods | 4 weeks
  postprandial systolic and diastolic blood pressure in mmHg at time 0
Changes in systolic and diastolic blood pressure at different postprandial periods | 4 weeks
  postprandial systolic and diastolic blood pressure in mmHg at 30 min
Changes in systolic and diastolic blood pressure at different postprandial periods | 4 weeks
  postprandial systolic and diastolic blood pressure in mmHg at 60 min
Changes in systolic and diastolic blood pressure at different postprandial periods | 4 weeks
  postprandial systolic and diastolic blood pressure in mmHg at 90 min
Changes in systolic and diastolic blood pressure at different postprandial periods | 4 weeks
  postprandial systolic and diastolic blood pressure in mmHg at 120 min

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriel Betanzos-Cabrera, Pachuca, Hidalgo, Mexico